CLINICAL TRIAL: NCT04966455
Title: Effect of Supplementing the Diet With Raisins, a Food Rich in Polyphenols, on Cognitive Function in Healthy Older Adults, a Randomised Controlled Trial
Brief Title: Effect of Raisins on Cognitive Function in Healthy Older Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, José Ignacio Recio Rodriguez, PhD in Biosciences, Principal Investigator, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GRS 2381/A/21
Record Dates: First submitted 2021-07-01; First posted 2021-07-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Cognitive Dysfunction
Keywords: Cognitive dysfunction; Heart Disease Risk Factors; Vitis; Polyphenols; Clinical Trial
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): No intervention
- Experimental group (Experimental): Supplementation of 50 g daily of rainsins for 3 months
  Interventions: Dietary Supplement: Raisins

INTERVENTIONS:
Dietary Supplement: Raisins — Daily supplementation of 50 g of rainsins for 3 months
  Arms: Experimental group

SUMMARY:
Objective:To assess the effect of an intervention based on including 50 g of raisins (sultanas) daily in the diet for 3 months on improving cognitive performance, cardiovascular risk factors and inflammatory markers in a population of older adults without cognitive impairment.

Methodology: Randomised two parallel-group clinical trial. Population: 80 patients between 70 and 80 years of age will be included, selected from primary care clinics in Salamanca and Zamora.

Measurements and intervention: Participants included in the study will have a baseline visit and two evaluations visits at 3 and 6 months where cognitive performance (attention, executive functions, verbal memory, working memory and language) will be assessed using a brief neuropsychological battery; quality of life, using the WHOQol- AGE and EUROQOL-5D questionnaire; blood pressure; glycaemia; body composition, using an impedancemeter; and different markers of inflammation, interleukin (IL) 6, IL-1 and tumour necrosis factor alpha (TNF); and different markers of inflammation, interleukin (IL) 6, IL-1 and tumour necrosis factor alpha (TNF-α).

Participants will be randomised using the Epidat 4.0 programme into 2 groups (control group and intervention group) with a ratio of 1:1. Both groups will be instructed to continue with their usual dietary pattern without changing their habits during the study period.

Those in the control group will not receive any amount of raisins to their usual diet. The participants in the intervention group will receive 50 g of raisins and instructions on the time of day to take it (at night). The duration of this intervention will be 3 months. The daily nutritional intake of this amount of raisins is as follows: 146 kcal; 0.25 g of fat; 34 g carbohydrates of which 34 g sugars; 1.3 g protein; 1 g fibre. The total polyphenol content of total polyphenols from 50 g of raisinas is approximately 532,5 mg (phenols explorer database).

ELIGIBILITY:
Inclusion Criteria:

* People of both sexes aged between 70 and 80 years.
* The score on the Mini Mental State Examination (MMSE) must be greater than or equal to 24 points.
* Self-employed to attend the centre where the study is carried out.
* Signature of the informed consent form.

Exclusion Criteria:

* Coronary or cerebrovascular atherosclerotic pathology.
* Diabetes mellitus
* Grade II or higher heart failure.
* Moderate or severe chronic obstructive pulmonary disease.
* Advanced renal or hepatic disease.
* Severe mental illness.
* Oncological disease under treatment diagnosed within the last 5 years or terminal condition.
* Morbid obesity (IMC ≥ 40 kg/m2).
* Intolerance and/or allergy to any of the grape components.
* Any other circumstance at the criterion of the researchers.

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-04-20 (Actual); Study Completion 2023-05-20 (Actual)

PRIMARY OUTCOMES:
Cognitive impairment | 3 months
  Evaluated by Montreal Cognitive Assessment (MoCA). Score (0-30). 30 (better score)

SECONDARY OUTCOMES:
Health-related quality of life | 3 months
  Evaluated by EuroQoL-5D-3L (EuroQol Visual Analogue Scale (EQ-VAS)) Range 0-100. 100 (best quality of life)
Health-related quality of life | 3 months
  Evaluated by EuroQoL-5D-3L (EQ-5D summary index ) Range 0-1. 1 (best quality of life)
Health-related quality of life | 3 months
  Evaluated by WHOQOL-AGE. Total score Range 0-65. 65 (best quality of life)
Blood pressure | 3 months
  Measured in mmHg
Plasma cholesterol | 3 months
  Measured in mg/dL
Inflammatory marker (IL-6 | 3 months
  Measured in pg/ml

CONTACTS AND LOCATIONS:
Overall Officials: Jose I Recio-Rodriguez, PhD, Principal Investigator — University of Salamanca
Locations (1):
- José Ignacio Recio Rodriguez, Salamanca, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rodrigo-Gonzalo MJ, Recio-Rodriguez JI, Mendez-Sanchez R, Pablos-Hernandez MC, Gonzalez-Ramirez A, Gonzalez-Sanchez J, Fermoso-Palmero MJ, Puente-Gonzalez AS, Sanchez-Sanchez MC, Barbero-Iglesias FJ, Rihuete-Galve MI, Gonzalez-Manzano S. Effect of including a dietary supplement of raisins, a food rich in polyphenols, on cognitive function in healthy older adults; a study protocol for a randomized clinical trial. BMC Geriatr. 2023 Mar 29;23(1):182. doi: 10.1186/s12877-023-03882-6. PMID 36991396